CLINICAL TRIAL: NCT04106830
Title: Prospective Cohort Study of CLinical and Imaging Patterns of NeUroinflammation DisEases (CLUE)
Brief Title: Clinical and Imaging Cohort of Neuroinflammation Diseases in China (CLUE)
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yaou Liu, Professor, Beijing Tiantan Hospital
Other Study IDs: KY2024-309-04
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: NMO Spectrum Disorder; MRI; Multiple Sclerosis; MOGAD
MeSH Terms: conditions — Neuromyelitis Optica; Multiple Sclerosis; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease | interventions — Azathioprine; Mycophenolic Acid; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- NMOSD: Patients with neuromyelitis optica spectrum disorders
  Interventions: Drug: Intravenous steroid
- Multiple sclerosis(MS): Patients with multiple sclerosis
  Interventions: Drug: Intravenous steroid
- MOGAD: Patients with myelin oligodendrocyte glycoprotein antibody-associated disease
  Interventions: Drug: Intravenous steroid
- Healthy controls (HC): Healthy people without any neuroinflammation disease

INTERVENTIONS:
Drug: Intravenous steroid — This study does not limit treatment methods.patients commonly use high-dose intravenous steroid therapy (HD-S) during acute stage. The HD-S treatment course referred to intravenous administration of 1 g of glucocorticoid daily for 3 consecutive days and continuous dose 240 mg reduction for 60mg oral administration. Immunomodulatory therapies are necessary for the remission stage. The treatment methods include: Azathioprine (start at 50 mg per day, add 50 mg per week to 2 mg/kg.d); Mycophenolate Mofetil (The initial dose was 0.25g bid, add 0.5g per week to 0.75g bid); and Rituximab (500 mg on the 1st day, the 15th day, then 500mg per half year).
  Other Names: Azathioprine; Mycophenolate Mofetil; Rituximab
  Groups: MOGAD; Multiple sclerosis(MS); NMOSD

SUMMARY:
CLUE is a prospective study to determine structural and functional changes of brain and spinal cord, as well as the inflammatory environment in patients with neuroinflammatory and demyelination disease. Participants will receive new magnetic resonance (MR) technics including double inversion recovery (DIR) imaging diffusion kurtosis imaging (DKI), quantitative susceptibility mapping (QSM) and resting-state functional imaging and follow up for one year using 3T MRI. In addition, participants will receive T1WI, T2WI, FLAIR and SWI sequences on 7T MRI.

DETAILED DESCRIPTION:
The study is an observational study of multi-model imaging to determine structural and functional changes of the brain, spinal cord and optic nervethe and inflammatory environment in patients with neuroinflammatory and demyelination disease. Brain, spinal cord and optic nerve involvement are common in neuroinflammatory and demyelination disease including clinical isolated syndrome (CIS), multiple sclerosis (MS), neuromyelitis optica spectrum disorders (NMOSDs), myelin oligodendrocyte glycoprotein antibody - associated disorders (MOGAD). The pathophysiology in neuroinflammatory disease involves the intensive autoimmune inflammatory response, resulting in demyelination and neuroaxonal injury and loss. Some cerebrospinal fluid (CSF) biomarkers have been reported to indicate the pathology and reflect disease activity, especially during the acute stage. However, they couldn't directly reflect the macroscopic and microscopic neuroaxonal change in the brain and spinal cord, which seem to be important determinants of long-term severe disability in chronic neuroinflammatory disease.

Finally, new MRI techniques are the most reliable and non-invasive method to assess the structure and function of brain and spinal cord, plus to monitor disease activity in clinical practice. Double inversion recovery (DIR) imaging allows better detection of cortical and white matter lesion, which has highlighted the role in MS. Diffusion kurtosis imaging (DKI) which has been proposed to characterize the deviation of water diffusion in neural tissues from Gaussian diffusion, is promising to provide information of demyelination and subsequent inflammatory processes in brain or spinal cord. Quantitative susceptibility mapping (QSM) has enabled MRI of tissue magnetic susceptibility to advance from simple qualitative detection of hypointense blooming artifacts to precise quantitative measurement of spatial biodistributions. QSM better depicts spatial susceptibility patterns in MS lesions compared to phase-based imaging. Besides, resting-state functional imaging has the potential to map the intrinsic functional brain networks and to detect early functional brain changes in neuroinflammatory disease.

This study will be a prospective cohort study of patients with neuroinflammatory and demyelination disease. Subjects will undertake MR scans at the acute stage and required follow-up visits after 1 month, 6 months, and 1 year. The MR scans are necessary at each visit.

This study does not limit treatment methods. Patients commonly use high-dose intravenous steroid therapy (HD-S) during the acute stage. The HD-S treatment course referred to intravenous administration of 1 g of glucocorticoid daily for 3 consecutive days and continuous dose 240 mg reduction for 60mg oral administration. Immunomodulatory therapies are necessary for the remission stage. The treatment methods include: Azathioprine (start at 50 mg per day, add 50 mg per week to 2 mg/kg*d); Mycophenolate Mofetil (The initial dose was 0.25g bid, add 0.5g per week to 0.75g bid); and Rituximab (500 mg on the 1st day, the 15th day, then 500mg per half year).

ELIGIBILITY:
Inclusion Criteria:

* 16-75
* Diagnosis of neuroinflammatory and demyelination disease
* Availability of demographic and clinical data at the time disease onset
* Informed written consent obtained from the patient, and/or patient's parent(s), and/or legal representative. Assent, if old enough to grant, will be obtained from all patients under the age of 16 years.

Exclusion Criteria:

* Patients for whom MRI is contra-indicated
* Patients included in an ongoing clinical trial where the product is blinded

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: To reflect the daily practices, this study includes all patients with neuroinflammatory and demyelination disease at the beginning of the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The brain structural change over time between the baseline MRI and the follow-up MRIs | On admission to the hospital on day 1, on discharge 180 days later and on follow up 360 days later
  To describe changes of lesions, grey matter and white matter in patients with neuroinflammatory and demyelination disease measured by DIR and QSM. The primary endpoint is the change over time between the baseline MRI and the follow-up MRIs, of the lesions and brain volumes.
The spinal cord change over time between the baseline MRI and the follow-up MRIs. | On admission to the hospital on day 1, on discharge 180 days later and on follow up 360 days later
  To describe changes of lesions and integrity of fiber bundle in spinal cord in neuroinflammatory and demyelination disease patients measured by DKI. The primary endpoint is the change over time between the baseline MRI and the follow-up MRIs, of structural change in spinal cord.
The functional change over time between the baseline MRI and the follow-up MRIs. | On admission to the hospital on day 1, on discharge 180 days later and on follow up 360 days later
  To describe brain functional changes in patients with neuroinflammatory and demyelination disease measured by resting-state functional imaging. The primary endpoint is the functional change over time between the baseline MRI and the follow-up MRIs

SECONDARY OUTCOMES:
Change from Baseline Expanded Disability Status Scale （EDSS）/ Functional Systems （FS） | On admission to the hospital on day 1, on discharge 180 days later and on follow up 360 days later
  admission to the hospital on day 1, on discharge 180 days later and on follow up 360 days later.] The Kurtzke Expanded Disability Status Scale (EDSS) was developed to measure the disability status of subjects with multiple sclerosis. It allows an objective quantification of the level of functioning that could be widely and reproducibly used by researchers and health care providers. The EDSS provides a total score on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability. The range of main categories include (0) = normal neurologic exam; to (5) = ambulatory without aid or rest for 200 meters; disability severe enough to impair full daily activities; to (10) = death due to Multiple sclerosis (MS). In addition, it also provides eight subscale measurements called Functional System (FS) scores.
Timed 25-foot Walk | On admission to the hospital on day 1, on discharge 180 days later and on follow up 360 days later
  Timed 25-foot walking trials will be assessed on admission to the hospital on day 1, on discharge 180 days later and on follow up 360 days later. The Timed 25-Foot Walk test is a quantitative measure of lower extremity function. If required, the subject may use an appropriate assistive device to walk as quickly as he/she can from one end to the other end of a clearly marked, unobstructed, 25-foot course. Timing will begin when any part of the subject's foot crosses the tape. Timing will end when any part of the subject's foot crosses the finish line (identified by a taped mark on the floor). Time will be recorded in seconds. The task is immediately administered again (a maximum five-minute rest period is allowed between trials) by having the subject walk back the same distance. The average of the two values will be recorded.
Mean change in visual acuity as assessed by Sloan 2.5% low contrast visual acuity chart. | On admission to the hospital on day 1, on discharge 180 days later and on follow up 360 days later
  admission to the hospital on day 1, on discharge 180 days later and on follow up 360 days later.] Low Contrast Visual Acuity: Low-contrast Sloan letter charts are readily available and provide a practical, quantitative, and standardized assessment of visual function. Each chart consists of rows of black letters (decreasing in size from top to bottom) on a white background.
  For this trial, 2.5% low contrast visual acuity will be measured on days 1 and 5 during the steroid phase and completion after the plasma exchange phase. Charts will be read at a 2.5-meter distance by trained examiners in the hospital room with constant lighting.

CONTACTS AND LOCATIONS:
Overall Officials: Yaou Liu, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Clinical and MR data can be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 5 years after the end of the trial.
Access Criteria: Neurologist and radiologist who submitting an application to Prof. Liu.

REFERENCES:
- [Derived] Xu Y, Ren Y, Li X, Xu W, Wang X, Duan Y, Liu Y, Zhang X, Tian DC. Persistently Gadolinium-Enhancing Lesion Is a Predictor of Poor Prognosis in NMOSD Attack: a Clinical Trial. Neurotherapeutics. 2021 Apr;18(2):868-877. doi: 10.1007/s13311-020-00973-9. Epub 2021 Jan 19. PMID 33469828